CLINICAL TRIAL: NCT02175121
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel Group Trial To Assess The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Multiple Oral Doses Of Pf-06291874 Given As Monotherapy To Adults With Type 2 Diabetes Mellitus
Brief Title: Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Study Of PF-06291874 As Oral Monotherapy To Treat Adults With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B4801011
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — PF-06291874

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Treatment B- PF-06291874 (Experimental)
  Interventions: Drug: PF-06291874
- Treatment C- PF-06291874 (Experimental)
  Interventions: Drug: PF-06291874
- Treatment D- PF-06291874 (Experimental)
  Interventions: Drug: PF-06291874
- Treatment E- PF-06291874 (Experimental)
  Interventions: Drug: PF-06291874

INTERVENTIONS:
Drug: Placebo — Tablet, once daily for 28 days
  Arms: Treatment A- Placebo
Drug: PF-06291874 — Tablet, 15 mg, once daily for 28 days
  Arms: Treatment B- PF-06291874
Drug: PF-06291874 — Tablet, 35 mg, once daily for 28 days
  Arms: Treatment C- PF-06291874
Drug: PF-06291874 — Tablet, 75 mg, once daily for 28 days
  Arms: Treatment D- PF-06291874
Drug: PF-06291874 — Tablet, 150 mg, once daily for 28 days
  Arms: Treatment E- PF-06291874

SUMMARY:
This study is going to assess the safety and tolerability of PF-06291874 in adults with Type 2 Diabetes Mellitus as monotherapy, to evaluate the significance of overall glycemic control in these subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects and non-childbearing potential female subjects between the ages of 18 and 70 years old.
* Body Mass Index of 18.0 to 45.4 kg/m2; and a total body weight of >50 kg
* HbA1c value at the screening visit meeting once of the following criteria:

  * Currently taking acceptable oral antiglycemic drug therapy within 6.5 to 9.5%
  * Not currently taking any oral antiglycemic drug therapy within 7 to 10.5%
* Fasting plasma glucose concentrations<270mg/dL at the screening and run-in visit, confirmed by a single repeat, if deemed necessary.
* Subjects must be willing and able to perform self-tests of blood glucose at least 4 times per day, and maintain a diary for the duration of participation in the study; and therefore, subjects must be literate.

Exclusion Criteria:

* History of Type 1 diabetes mellitus or secondary forms of diabetes
* One or more self-reported hypoglycemic episodes of sever intensity within 3 months of screening; or 2 or more self-reported hypoglycemic episodes of severe intensity within the previous 6 months.
* History of myocardial infarction, unstable angina, arterial revascularization, stroke, New York Heart Association Functional Class II-IV heart failure, or transient ischemic attach within 6 months of screening.
* History or evidence of diabetic complications with significant end organ damage, such as

  * Proliferative retinopathy and/or macular edema;
  * Diabetic neuropathy complicated by neuropathic ulcers;
* Screening seated systolic blood pressure >160 mm Hg and/or diastolic blood pressure >100 mm Hg after at least a 5 minute seated rest. If the blood pressure exceeds this limit, the blood pressure may be repeated 2 more times following approximately 2 minutes of rest between measurements and the median of the 3 values should be used to determine subject eligibility;
* Male subjects with partners currently pregnant; or male subjects capable of conceiving children who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (18):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Profil Institute for Clinical Research, Inc., Chula Vista, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - SeaView Research, Inc., Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - Miami Research Associates, Inc., South Miami, Florida
  - MRA Clinical Research, LLC, South Miami, Florida
  - MRA Clinical Research, South Miami, Florida
  - Louisville Metabolic and Atherosclerosis Research Center, Louisville, Kentucky
  - DaVita Clinical Research, Minneapolis, Minnesota
  - Clinilabs, Inc., Eatontown, New Jersey
  - PRA International, Marlton, New Jersey
  - Buffalo Clinical Research Center, LLC, Buffalo, New York
  - High Point Clinical Trials Center, LLC, High Point, North Carolina
  - Community Research, Cincinnati, Ohio
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Rainier Clinical Research Center, Inc., Renton, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4801011&StudyName=Safety%2C%20Tolerability%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Study%20Of%20PF-06291874%20As%20Oral%20Monotherapy%20To%20Treat%20Adults%20With%20Type%202%20Diabete

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligibility included male participants or female participants of non-childbearing potential, 18 to 70 years of age (inclusive) who were willing and able to wash off all diabetes medications.
Groups:
- Placebo: Participants received placebo (three 5/25 milligram [mg] and one 100 mg matching placebo tablets) once daily for 28 days
- PF-06291874 15 mg: Participants received PF-06291874 15 mg (three 5 mg tablets and one 100 mg placebo tablet) once daily for 28 days
- PF-06291874 35 mg: Participants received PF-06291874 35 mg (two 5 mg tablets, one 25 mg tablet and one 100 mg placebo tablet) once daily for 28 days
- PF-06291874 75 mg: Participants received PF-06291874 75 mg (three 25 mg tablets and one 100 mg placebo tablet) once daily for 28 days
- PF-06291874 150 mg: Participants received PF-06291874 150 mg (two 25 mg tablets, one 100 mg tablet and one 5/25 mg placebo tablet) once daily for 28 days
Period: Overall Study
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Started | 34 | 35 | 34 | 35 | 34
Completed | 33 | 34 | 32 | 34 | 33
Not Completed | 1 | 1 | 2 | 1 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0
Not completed — Personal emergency | 0 | 0 | 0 | 0 | 1
Not completed — Schedule conflict | 0 | 0 | 1 | 0 | 0
Not completed — Time issues | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg | Total
Number analyzed (Participants) | 34 | 35 | 34 | 35 | 34 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (6.3) | 56.1 (9) | 57.8 (7.5) | 55.5 (7.6) | 55.2 (7.5) | 56.7 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 16 | 12 | 18 | 71
  Male | 18 | 26 | 18 | 23 | 16 | 101

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), or Serious Adverse Events (SAEs), or Hypoglycemic Adverse Events (HAE) or Withdrawals Due to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life threatening (immediate risk of death); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. An HAE was identified by characteristic symptoms or blood glucose levels. TEAEs are events between first dose of study drug and up to 10-14 days after last dose of study drug that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline up to 10-14 days after last dose of study drug, up to 42 days
Population: The safety analysis set was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 34 | 35 | 34 | 35 | 34
participants
  Number of Participants With AEs | 11 | 7 | 10 | 11 | 12
  Number of Participants with SAEs | 0 | 0 | 0 | 1 | 0
  Number of Participants with Protocol-Defined HAEs | 0 | 0 | 0 | 1 | 0
  Number of Participants discontinued from study | 1 | 1 | 2 | 1 | 1

2. Primary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: The total number of participants with laboratory test abnormalities (without regard to baseline abnormality) was assessed. Clinical laboratory tests included hematology, chemistry, urinalysis, and some other tests.
Time Frame: Baseline up to 10-14 days after last dose of study drug, up to 42 days
Population: The safety analysis set was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 34 | 35 | 34 | 35 | 34
participants | 31 | 31 | 24 | 32 | 30

3. Primary Outcome: Number of Participants With Change From Baseline and Absolute Values in Vital Signs Meeting Criteria of Potential Clinical Concern
Description: Vital Signs included seated supine systolic and diastolic blood pressure (BP) and pulse rate. Vital signs criteria of potential clinical concern were 1), BP: systolic (SBP) greater than or equal to (>=) 30 millimeters of mercury (mm Hg) change from baseline, systolic less than (<) 90 mm Hg; diastolic BP (DBP) >=20 mm Hg change from baseline, diastolic <50 mm Hg; 2), pulse rate <40 or greater than (>) 120 beats per minute (bpm).
Time Frame: Baseline up to 10-14 days after last dose of study drug, up to 42 days
Population: The safety analysis set was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 34 | 35 | 34 | 35 | 34
participants
  Supine SBP <90 mm Hg | 3 | 0 | 0 | 0 | 0
  Supine DBP <50 mm Hg | 1 | 0 | 0 | 0 | 0
  Increase: supine SBP >=30 mm Hg | 3 | 3 | 3 | 1 | 6
  Increase: supine DBP >=20 mm Hg | 1 | 0 | 2 | 1 | 0
  Decrease: supine SBP >= 30 mm Hg | 1 | 0 | 0 | 0 | 0
  Decrease: supine DBP >=20 mm Hg | 3 | 0 | 0 | 0 | 0
  Pulse rate <40 bpm | 0 | 0 | 0 | 0 | 0
  Pulse rate >120 bpm | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Criteria of Potential Clinical Concern
Description: ECG criteria of potential clinical concern were 1), time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization (QRS interval): >=140 msec; >=50% increase from baseline; 2), the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization (PR interval): >=300 milliseconds (msec); >=25 percent (%) increase when baseline >200 msec; or increase >=50% when baseline less than or equal to (<=)200 msec; 3), time from ECG Q wave to the end of the T wave corresponding to electrical systole corrected for heart rate using Fridericia's formula (QTcF interval): absolute value >=450 - <480 msec, >=480-<500 msec, >=500 msec; increase from baseline >=30 - <60, >=60 msec.
Time Frame: Baseline up to 10-14 days after last dose of study drug, up to 42 days
Population: The safety analysis set was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 34 | 35 | 34 | 35 | 34
participants
  PR interval >=300 msec | 0 | 0 | 0 | 0 | 0
  QRS interval >=140 msec | 0 | 0 | 0 | 0 | 0
  QTcF interval 450-480 msec | 2 | 4 | 4 | 2 | 3
  QTcF interval 480-500 msec | 0 | 0 | 1 | 0 | 1
  QTcF interval >=500 msec | 0 | 0 | 0 | 0 | 0
  PR interval increase >=25%/50% | 0 | 1 | 0 | 0 | 0
  QRS interval increase >=50% | 0 | 0 | 0 | 0 | 0
  QTcF interval increase 30-60 msec | 1 | 5 | 4 | 4 | 5
  QTcF interval increase >=60 msec | 0 | 0 | 1 | 0 | 0

5. Secondary Outcome: Change From Baseline in Mean Daily Glucose
Description: The mean daily glucose was determined from the area under the concentration (AUC) of the glucose concentrations measured at nominal times 0, 0.5, 1, 1.5, 2, 4, 6, 10, 12, 15 and 24 hours post dose. Mean daily glucose change from baseline (defined as Day 0) on Day 28.
Time Frame: Baseline and Day 28
Population: The full analysis set (FAS) was used in the analysis of the pharmacodynamic (PD) parameters. The FAS was defined as all subjects randomized and who received at least 1 dose of randomized treatment. Number of participants analyzed represents the available number of participants for analysis at post-baseline days.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 33 | 35 | 31 | 35 | 33
mg/dL | 6.63 (38.938) [2.33 to 18.37] | -29.15 (25.659) [-37.73 to -22.22] | -32.29 (29.572) [-43.44 to -26.93] | -59.98 (29.363) [-66.19 to -50.68] | -55.99 (39.798) [-65.76 to -49.78]
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p < 0.0001, ANCOVA — Two-sided p-values are from analysis of Covariance (ANCOVA) model with baseline value and treatment group as fixed effects; LS mean difference from placebo adjusted for baseline values is derived from the ANCOVA model; Mean Difference (Net) = -40.33, 90% CI 2-sided [-51.49 to -29.16], Standard Error of Mean 6.75
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 35 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference from placebo adjusted for baseline values is derived from the ANCOVA model; Mean Difference (Net) = -45.53, 90% CI 2-sided [-57.08 to -33.99], Standard Error of Mean 6.98
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 75 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference from placebo adjusted for baseline values is derived from the ANCOVA model; Mean Difference (Net) = -68.79, 90% CI 2-sided [-79.92 to -57.65], Standard Error of Mean 6.73
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference from placebo adjusted for baseline values is derived from the ANCOVA model; Mean Difference (Net) = -68.12, 90% CI 2-sided [-79.46 to -56.78], Standard Error of Mean 6.86

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: Fasting plasma glucose response change from baseline (defined as the mean of Day 0 and Day 1 pre-dose) on Day 14, and the mean of Days 28 and 29.
Time Frame: Baseline, Day 14 and the mean of Days 28 and 29
Population: The FAS was used in the analysis of the PD parameters. The FAS was defined as all subjects randomized and who received at least 1 dose of randomized treatment. N in change from Baseline when different, represents the available number of participants for analysis at post-baseline days.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 34 | 35 | 34 | 35 | 34
mg/dL
  Day 14 Change from Baseline (N=33,34,32,35,33) | -6.08 (29.778) | -21.76 (24.278) | -29.59 (31.552) | -45.59 (26.040) | -52.18 (30.824)
  Day 28 Change from Baseline (N=33,35,32,35,33) | 6.11 (29.840) | -20.26 (23.523) | -26.61 (22.045) | -45.27 (22.115) | -50.45 (32.045)
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.0060, Mixed Models Analysis — Two-sided p-values are from MMRM with baseline value, time, treatment group, study day and treatment interaction as fixed effects. Subject was used as a random effect; Mean Difference (Net) = -16.25, 90% CI 2-sided [-25.90 to -6.60], Standard Error of Mean 5.83
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 35 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Net) = -26.98, 90% CI 2-sided [-36.81 to -17.15], Standard Error of Mean 5.94
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 75 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Net) = -39.60, 90% CI 2-sided [-49.20 to -30.00], Standard Error of Mean 5.80
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Net) = -46.72, 90% CI 2-sided [-56.46 to -36.98], Standard Error of Mean 5.89
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Net) = -27.07, 90% CI 2-sided [-35.89 to -18.25], Standard Error of Mean 5.33
Statistical Analysis 6: Comparison: Placebo vs PF-06291874 35 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Net) = -36.18, 90% CI 2-sided [-45.21 to -27.14], Standard Error of Mean 5.46
Statistical Analysis 7: Comparison: Placebo vs PF-06291874 75 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Net) = -51.47, 90% CI 2-sided [-60.29 to -42.65], Standard Error of Mean 5.33
Statistical Analysis 8: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Net) = -57.17, 90% CI 2-sided [-66.12 to -48.22], Standard Error of Mean 5.41

7. Secondary Outcome: Percent Change From Baseline in Triglycerides
Description: Triglycerides percent change from baseline (defined as the mean of Day 0 and Day 1 pre-dose) on Day 14, and the mean of Days 28 and 29.
Time Frame: Baseline, Day 14 and the mean of Days 28 and 29
Population: The FAS was used in the analysis of the PD parameters. The FAS was defined as all subjects randomized and who received at least 1 dose of randomized treatment. N in percent change from Baseline when different, represents the available number of participants for analysis at post-baseline days.
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 34 | 35 | 34 | 35 | 34
% (percent change)
  D14 Percent Change from Baseline(N=33,35,32,35,33) | 0.52 (47.749) | 25.69 (93.991) | 26.95 (100.972) | 2.71 (63.990) | 21.52 (86.951)
  D28 Percent Change from Baseline(N=33,35,32,35,33） | 19.58 (26.037) | 15.20 (29.122) | 19.48 (28.647) | 20.72 (40.626) | 24.96 (35.090)
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.2063, Mixed Models Analysis — Two-sided p-values are from MMRM with baseline value, time, treatment group, study day, statin use and treatment interaction as fixed effects. Subject was used as a random effect; Mean Difference (Net) = 12.86, 90% CI 2-sided [-3.91 to 29.62], Standard Error of Mean 10.13
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 35 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.2087, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 13.03, 90% CI 2-sided [-4.05 to 30.11], Standard Error of Mean 10.33
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 75 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.5802, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 5.60, 90% CI 2-sided [-11.11 to 22.30], Standard Error of Mean 10.10
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.1553, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 14.64, 90% CI 2-sided [-2.32 to 31.59], Standard Error of Mean 10.25
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.7741, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -2.20, 90% CI 2-sided [-14.87 to 10.47], Standard Error of Mean 7.66
Statistical Analysis 6: Comparison: Placebo vs PF-06291874 35 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.9588, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -0.40, 90% CI 2-sided [-13.28 to 12.47], Standard Error of Mean 7.78
Statistical Analysis 7: Comparison: Placebo vs PF-06291874 75 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.8523, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 1.42, 90% CI 2-sided [-11.17 to 14.01], Standard Error of Mean 7.61
Statistical Analysis 8: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.4166, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 6.30, 90% CI 2-sided [-6.49 to 19.08], Standard Error of Mean 7.73

8. Secondary Outcome: Percent Change From Baseline in Total Cholesterol
Description: Total cholesterol percent change from baseline (defined as the mean of Day 0 and Day 1 pre-dose) on Day 14, and the mean of Days 28 and 29.
Time Frame: Baseline, Day 14 and the mean of Days 28 and 29
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 34 | 35 | 34 | 35 | 34
% (percent change)
  D14 Percent Change from Baseline(N=33,35,32,35,33) | 4.04 (11.024) | 4.49 (11.036) | 7.94 (16.059) | 4.60 (12.888) | 12.98 (17.177)
  D28 Percent Change from Baseline(N=33,35,32,35,33) | 4.07 (7.928) | 2.93 (11.503) | 4.52 (11.354) | 4.05 (13.061) | 12.86 (17.086)
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.8516, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 0.60, 90% CI 2-sided [-4.73 to 5.93], Standard Error of Mean 3.22
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 35 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.2303, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 3.97, 90% CI 2-sided [-1.48 to 9.42], Standard Error of Mean 3.29
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 75 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.7132, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 1.19, 90% CI 2-sided [-4.15 to 6.52], Standard Error of Mean 3.22
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.0034, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 9.74, 90% CI 2-sided [4.32 to 15.16], Standard Error of Mean 3.28
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.7394, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -0.99, 90% CI 2-sided [-5.89 to 3.92], Standard Error of Mean 2.96
Statistical Analysis 6: Comparison: Placebo vs PF-06291874 35 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.8652, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 0.52, 90% CI 2-sided [-4.50 to 5.53], Standard Error of Mean 3.03
Statistical Analysis 7: Comparison: Placebo vs PF-06291874 75 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.8370, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 0.61, 90% CI 2-sided [-4.30 to 5.52], Standard Error of Mean 2.97
Statistical Analysis 8: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.0018, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 9.59, 90% CI 2-sided [4.60 to 14.58], Standard Error of Mean 3.01

9. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein-Cholesterol (LDL-C)
Description: LDL-C percent change from baseline (defined as the mean of Day 0 and Day 1 pre-dose) on Day 14, and the mean of Days 28 and 29.
Time Frame: Baseline, Day 14 and the mean of Days 28 and 29
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 34 | 35 | 34 | 35 | 34
% (percent change)
  D14 Percent Change from Baseline(N=33,35,32,35,33) | 6.24 (15.803) | 3.95 (14.407) | 8.12 (23.085) | 5.29 (15.223) | 14.24 (21.612)
  D28 Percent Change from Baseline(N=33,35,32,35,33) | 2.92 (12.046) | 2.46 (13.472) | 3.51 (19.507) | 2.15 (17.238) | 14.19 (24.128)
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.6182, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -2.12, 90% CI 2-sided [-9.15 to 4.91], Standard Error of Mean 4.25
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 35 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.7028, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 1.66, 90% CI 2-sided [-5.52 to 8.84], Standard Error of Mean 4.34
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 75 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.9445, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -0.30, 90% CI 2-sided [-7.33 to 6.73], Standard Error of Mean 4.25
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.0373, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 9.07, 90% CI 2-sided [1.93 to 16.21], Standard Error of Mean 4.32
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.9448, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -0.29, 90% CI 2-sided [-7.25 to 6.67], Standard Error of Mean 4.21
Statistical Analysis 6: Comparison: Placebo vs PF-06291874 35 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.9312, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 0.37, 90% CI 2-sided [-6.74 to 7.49], Standard Error of Mean 4.30
Statistical Analysis 7: Comparison: Placebo vs PF-06291874 75 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.9791, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -0.11, 90% CI 2-sided [-7.07 to 6.85], Standard Error of Mean 4.21
Statistical Analysis 8: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.0044, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 12.34, 90% CI 2-sided [5.26 to 19.41], Standard Error of Mean 4.28

10. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein-Cholesterol (HDL-C)
Description: HDL-C percent change from baseline (defined as the mean of Day 0 and Day 1 pre-dose) on Day 14, and the mean of Days 28 and 29.
Time Frame: Baseline, Day 14 and the mean of Days 28 and 29
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 34 | 35 | 34 | 35 | 34
% (percent change)
  D14 Percent Change from Baseline(N=33,35,32,35,33) | 6.99 (15.590) | 9.02 (14.884) | 11.27 (15.720) | 14.47 (16.884) | 19.75 (18.172)
  D28 Percent Change from Baseline(N=33,35,32,35,33) | 3.94 (11.330) | 4.78 (9.271) | 4.82 (13.426) | 8.34 (9.013) | 18.73 (24.979)
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.6553, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 1.77, 90% CI 2-sided [-4.78 to 8.33], Standard Error of Mean 3.96
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 35 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.2569, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 4.61, 90% CI 2-sided [-2.09 to 11.30], Standard Error of Mean 4.05
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 75 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.0553, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 7.64, 90% CI 2-sided [1.09 to 14.18], Standard Error of Mean 3.96
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 12.89, 90% CI 2-sided [6.26 to 19.53], Standard Error of Mean 4.01
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.8717, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 0.58, 90% CI 2-sided [-5.35 to 6.51], Standard Error of Mean 3.58
Statistical Analysis 6: Comparison: Placebo vs PF-06291874 35 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.7430, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 1.20, 90% CI 2-sided [-4.86 to 7.26], Standard Error of Mean 3.66
Statistical Analysis 7: Comparison: Placebo vs PF-06291874 75 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.2041, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 4.56, 90% CI 2-sided [-1.36 to 10.48], Standard Error of Mean 3.58
Statistical Analysis 8: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 14.92, 90% CI 2-sided [8.92 to 20.92], Standard Error of Mean 3.63

11. Secondary Outcome: Percent Change From Baseline in Non-HDL-C
Description: Non-HDL-C percent change from baseline (defined as the mean of Day 0 and Day 1 pre-dose) on Day 14, and the mean of Days 28 and 29.
Time Frame: Baseline, Day 14 and the mean of Days 28 and 29
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 34 | 35 | 34 | 35 | 34
% (percent change)
  D14 Percent Change from Baseline(N=33,35,32,35,33) | 3.29 (11.686) | 2.96 (14.179) | 7.52 (20.983) | 1.26 (16.181) | 12.32 (22.192)
  D28 Percent Change from Baseline(N=33,35,32,35,33) | 3.84 (8.728) | 2.55 (14.319) | 4.65 (14.309) | 2.75 (17.275) | 12.32 (22.758)
Statistical Analysis 1: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.9750, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 0.13, 90% CI 2-sided [-6.62 to 6.87], Standard Error of Mean 4.08
Statistical Analysis 2: Comparison: Placebo vs PF-06291874 35 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.3396, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 3.99, 90% CI 2-sided [-2.90 to 10.87], Standard Error of Mean 4.16
Statistical Analysis 3: Comparison: Placebo vs PF-06291874 75 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.7142, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -1.49, 90% CI 2-sided [-8.23 to 5.24], Standard Error of Mean 4.07
Statistical Analysis 4: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test for Day 14; Test type: Superiority or Other; p = 0.0192, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 9.78, 90% CI 2-sided [2.94 to 16.63], Standard Error of Mean 4.14
Statistical Analysis 5: Comparison: Placebo vs PF-06291874 15 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.8277, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -0.84, 90% CI 2-sided [-7.20 to 5.52], Standard Error of Mean 3.85
Statistical Analysis 6: Comparison: Placebo vs PF-06291874 35 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.8857, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 0.57, 90% CI 2-sided [-5.93 to 7.06], Standard Error of Mean 3.93
Statistical Analysis 7: Comparison: Placebo vs PF-06291874 75 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.8824, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = -0.57, 90% CI 2-sided [-6.93 to 5.79], Standard Error of Mean 3.84
Statistical Analysis 8: Comparison: Placebo vs PF-06291874 150 mg; Placebo was the Reference and each of the active doses was the Test for Day 28; Test type: Superiority or Other; p = 0.0192, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Net) = 9.23, 90% CI 2-sided [2.77 to 15.69], Standard Error of Mean 3.90

12. Secondary Outcome: Percent Change From Baseline in Oxidized LDL
Description: Oxidized LDL percent change from baseline (defined as the mean of Day 0 and Day 1 pre-dose) on Day 28 (the mean of Days 28 and 29).
Time Frame: Baseline and the mean of Days 28 and 29
Population: The FAS was used in the analysis of the PD parameters. The FAS was defined as all subjects randomized and who received at least 1 dose of randomized treatment. Number of participants analyzed represents the available number of participants for analysis at post-baseline days.
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 33 | 35 | 32 | 35 | 33
% (percent change) | 2.84 (10.730) | 2.83 (13.474) | 6.54 (17.054) | 2.05 (16.179) | 11.93 (18.012)

13. Secondary Outcome: Percent Change From Baseline in Large LDL Particles
Description: Large LDL particles percent change from baseline (defined as the mean of Day 0 and Day 1 pre-dose) on Day 28 (the mean of Days 28 and 29).
Time Frame: Baseline and the mean of Days 28 and 29
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 32 | 35 | 31 | 35 | 33
% (percent change) | 3.49 (52.827) | 33.07 (116.700) | -2.40 (28.818) | -3.27 (37.299) | 21.49 (63.913)

14. Secondary Outcome: Percent Change From Baseline in Medium Small LDL Particles
Description: Medium small LDL particles percent change from baseline (defined as the mean of Day 0 and Day 1 pre-dose) on Day 28 (the mean of Days 28 and 29).
Time Frame: Baseline and the mean of Days 28 and 29
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 32 | 35 | 31 | 35 | 33
% (percent change) | 2.50 (34.138) | 8.19 (29.408) | 9.90 (35.164) | 8.32 (28.865) | 14.31 (35.623)

15. Secondary Outcome: Percent Change From Baseline in Small LDL Particles
Description: Small LDL particles percent change from baseline (defined as the mean of Day 0 and Day 1 pre-dose) on Day 28 (the mean of Days 28 and 29).
Time Frame: Baseline and the mean of Days 28 and 29
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 32 | 35 | 31 | 35 | 33
% (percent change) | 2.60 (32.581) | 7.58 (47.408) | 13.21 (42.540) | 3.67 (27.883) | 13.21 (38.033)

16. Secondary Outcome: Percent Change From Baseline in Very Small LDL Particles
Description: Very small LDL particles percent change from baseline (defined as the mean of Day 0 and Day 1 pre-dose) on Day 28 (the mean of Days 28 and 29).
Time Frame: Baseline and the mean of Days 28 and 29
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 32 | 35 | 31 | 35 | 33
% (percent change) | 2.87 (33.545) | 8.39 (57.323) | 14.25 (46.491) | 2.61 (28.176) | 12.92 (39.082)

17. Secondary Outcome: Percent Change From Baseline in Total LDL Particles
Description: Total LDL particles percent change from baseline (defined as the mean of Day 0 and Day 1 pre-dose) on Day 28 (the mean of Days 28 and 29).
Time Frame: Baseline and the mean of Days 28 and 29
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 32 | 35 | 31 | 35 | 33
% (percent change) | 1.33 (16.399) | 0.62 (13.142) | 3.39 (20.100) | 1.95 (17.192) | 13.70 (23.707)

18. Secondary Outcome: Percent Change From Baseline in LDL Size
Description: The LDL size percent change from baseline (defined as the mean of Day 0 and Day 1 pre-dose) on Day 28 (the mean of Days 28 and 29).
Time Frame: Baseline and the mean of Days 28 and 29
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 32 | 35 | 31 | 35 | 33
% (percent change) | -0.10 (2.294) | 0.16 (1.814) | -0.19 (1.604) | -0.26 (1.803) | 0.23 (2.018)

19. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B100
Description: The Apolipoprotein B100 was calculated as the difference between total Apolipoprotein B and Apolipoprotein B48 and analyzed the percent change from baseline (defined as mean of Day 0 and Day 1) on Day 28 (mean of Days 28 and 29).
Time Frame: Baseline and the mean of Days 28 and 29
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 33 | 35 | 32 | 35 | 33
% (percent change) | 1.85 (7.912) | 2.94 (11.436) | 3.82 (13.694) | 2.04 (13.900) | 10.35 (18.035)

20. Secondary Outcome: Percent Change From Baseline in Lipoprotein A
Description: The Lipoprotein A percent change from baseline (defined as the mean of Day 0 and Day 1 pre-dose) on Day 28 (mean of Days 28 and 29).
Time Frame: Baseline and the mean of Days 28 and 29
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: % (percent change)
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 33 | 35 | 32 | 35 | 33
% (percent change) | -4.38 (16.100) | -12.78 (15.095) | -13.48 (15.739) | -13.17 (16.639) | -15.15 (19.449)

21. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: Maximum PF-06291874 plasma concentration.
Time Frame: Day 28 (samples taken at 0, 2, 4, 8 and 24 hours after Day 28 dose)
Population: The PK analysis set was defined as all participants who received at least 1 dose of study medication. Samples for participants taking placebo were not analyzed. Number of participants analyzed represents the available number of participants for analysis at post-baseline days.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 35 | 31 | 35 | 33
ng/mL | 714.3 (25) | 1819 (29) | 3560 (28) | 8265 (27)

22. Secondary Outcome: Time to Reach Cmax (Tmax)
Description: Time to maximum PF-06291874 plasma concentration.
Time Frame: Day 28 (samples taken at 0, 2, 4, 8 and 24 hours after Day 28 dose)
Population: as for outcome 21
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 35 | 31 | 35 | 33
hour (hr) | 6.00 [2.00 to 8.02] | 6.00 [2.00 to 8.02] | 6.00 [2.00 to 24.0] | 6.00 [3.92 to 8.02]

23. Secondary Outcome: Area Under the Concentration-Time Profile From Zero to Time Tau (AUCtau) (Where Tau=24 Hours)
Description: Area under the PF-06291874 plasma concentration-time profile from time zero to time tau, the dosing interval, where tau=24 hours.
Time Frame: Day 28 (samples taken at 0, 2, 4, 8 and 24 hours after Day 28 dose)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 35 | 31 | 35 | 32
ng*hr/mL | 12760 (29) | 32370 (32) | 65230 (31) | 142900 (32)

24. Secondary Outcome: Minimum Plasma Concentration (Cmin)
Description: Minimum PF-06291874 plasma concentration.
Time Frame: Day 28 (samples taken at 0, 2, 4, 8 and 24 hours after Day 28 dose)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 35 | 31 | 35 | 32
ng/mL | 350.6 (46) | 666.4 (305) | 1257 (361) | 3247 (233)

25. Secondary Outcome: Apparent Clearance (CL/F)
Description: Apparent oral clearance of PF-06291874.
Time Frame: Day 28 (samples taken at 0, 2, 4, 8 and 24 hours after Day 28 dose)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Number analyzed (Participants) | 35 | 31 | 35 | 32
L/hr | 1.176 (29) | 1.082 (32) | 1.150 (31) | 1.050 (32)

ADVERSE EVENTS:
Time Frame: From Baseline to 10-14 days after the last dose of the study drug, up to 42 days
Arm/Group | Placebo | PF-06291874 15 mg | PF-06291874 35 mg | PF-06291874 75 mg | PF-06291874 150 mg
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35 | 0/34 | 1/35 | 0/34
Other Adverse Events (participants affected / at risk) | 4/34 | 4/35 | 8/34 | 6/35 | 6/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=34) | PF-06291874 15 mg (N=35) | PF-06291874 35 mg (N=34) | PF-06291874 75 mg (N=35) | PF-06291874 150 mg (N=34)
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=34) | PF-06291874 15 mg (N=35) | PF-06291874 35 mg (N=34) | PF-06291874 75 mg (N=35) | PF-06291874 150 mg (N=34)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 3 | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3
Fatigue (General disorders) | 0 | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 3 | 4 | 1
Headache (Nervous system disorders) | 1 | 0 | 3 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.